CLINICAL TRIAL: NCT02217371
Title: Role of Circadian and Homeostatic Systems in the Regulation of Wakefulness in Adult Patients With Attention Deficit Disorder With or Without Hyperactivity
Acronym: VEILLETDAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2013/06
Record Dates: First submitted 2014-05-05; First posted 2014-08-15 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: ADHD Patient; Healthy subjects; Sleepiness; PSG; MWT; EEG; cognitive tests
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Sleepiness | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADHD patient (Experimental)
  Interventions: Other: Neuropsychological tests
- Healthy volunteers (Active Comparator)
  Interventions: Other: Neuropsychological tests

INTERVENTIONS:
Other: Neuropsychological tests — The tests are :
  Go/NoGo paradigm, Continuous Performance Test (CPT) II , Wisconsin Card Sorting Test (WCST), virtual CPT, Classic and virtual Stroop, PSG, MWT
  These tests will be repeated during 32h each 4h (T0h, T4h, T8h, T12h, T16h, T20h, T24h, T28h et T32h).

SUMMARY:
In a previous protocol, we highlighted an excessive daytime sleepiness at the Maintenance of Wakefulness Tests (MWT) in 36% of adult Attention Deficit Disorder with or without Hyperactivity (ADHD) patients. In 40% of cases this sleepiness was associated with a sleep disorder objectified by polysomnography (PSG): apnea hypopnea syndrome (AHI) ≥ 10/h and / or Periodicals Movements of Lower Limb (PLMI) ≥ 15/h. However, among patients with no sleep disorder PSG, we can question the central origin of the Excessive Daytime Sleepiness. Thus, we wish to determine potential changes in the regulation of sleep / wake cycle through a protocol of extended wake.

The principal objective is to compare the objective sleepiness in sleepy patients with ADHD and healthy subjects during a protocol of extended wake.

It's an observational study of interventional type realized in patient with ADHD syndrome deprived of psychostimulant treatment (for 72 hours) and healthy subject, investigating the implication of the homeostatic and circadian systems in the preservation of awakening.

ELIGIBILITY:
Inclusion Criteria:

For ADHD patient:

* Patients male or feminine, from 18 to 50 years old,
* Patient respondent in the criterion current diagnosis of the ADHD according to the Diagnostic and Statistical Manual of Mental Disorders (DSM) IV-TR,
* Meeting the criteria diagnosis of ADHD in the childhood, estimated by the interview " Conners'Adult ADHD Diagnostic Interview for DSM-IV " (CAADID),
* Patient presenting a total score ≥ 20 at CAARS With at least 6 items of money scales inattention or hyperactivity ≥ 2,
* Patients deprived of any psychostimulants for 72 hours,
* Presenting at the polygraphy the absence of night-respiratory disorders (AHI < 10 / hour) and of Periodic Limbs Movements (PLMI < 15 / hour), as well as the absence of restless legs syndrome at the interview,
* Presenting to the MWT an excessive daytime sleepiness: mean latency < 20 min,
* Absence of syndrome of phase delay according to the criteria of l'ICSD2 (International Classification Sleep Disorders),
* Having been schooled until class of 3rd,
* Having regular schedules of life 4 days before going into the study,
* Beneficiary of a national insurance scheme,
* Having given in writing their informed consent to participate in the study.

For healthy subject:

* Patients male or feminine, from 18 to 50 years old,
* Subjects not symptomatic of ADHD (Total score at the Wender Utah Rating Scale strictly lower than 46 on 25 questions concerning the ADHD, and less than four crosses in the more darker cases of first 6 questions of ASRS),
* Subjects not presenting complaints of sleep, nor excessive daytime sleepiness (No item equal to 4 or 5 at Basic Nordic Sleep Questionnaire (BNSQ), excepted items 16 and 17 and total score at the Epworth Sleepiness Scale < 11),
* Presenting at the polygraphy the absence of night-respiratory disorders (AHI < 10 / hour) and of Periodic Limbs Movements (PLMI < 15 / hour), as well as the absence of restless legs syndromeat the interview,
* Not presenting to the MWT an excessive daytime sleepiness: mean latency > 34 min,
* Absence of syndrome of phase delay according to the criteria of l'ICSD2 (International Classification Sleep Disorders),
* Having been schooled until class of 3rd,
* Having regular schedules of life 4 days before going into the study,
* Beneficiary of a national insurance scheme,
* Having given in writing their informed consent to participate in the study.

Exclusion Criteria:

* Posted or night work,
* Any evolutionary affection (Brain tumour, epilepsy, migraine, cerebral vascular accident, calcifies, myoclonia, chorea, neuropathy, muscular dystrophies, dystrophy myotonic…),
* Psychiatric comorbidity: Current major depressive episode, current hypo obsessive or obsessive episode, schizophrenia,
* Renal disorders (Renal insufficiency, nephrolithiasis...),
* Endocrine pathologies (dysthyroidism, diabetes),
* Drug addiction during the last 6 months,
* Alcohol addiction during the last 6 months,
* Dependence in the tetra-hydroxy-cannabinol during the last 6 months,
* Long-term treatment by benzodiazepines,
* Treatment by atomoxetine,
* Pregnant and breast-feeding women,
* People under supervision, guardianship,
* Person incapable to give personally its consent,
* Nobody in emergency situation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Comparison of objective sleepiness | at inclusion (day 0)
  Comparison of objective sleepiness in sleepy patients with ADHD and healthy subjects during a protocol of extended wake.

SECONDARY OUTCOMES:
Theta-alpha band of EEG sleep | At inclusion (Day 0)
  Time constant and asymptotic value of the spectral power of the theta-alpha band of EEG sleep
Amplitude and phase of internal temperature | At inclusion (day 0)
Score of Karolinska Sleepiness Scale (subjective measure of sleepiness) | At inclusion (day 0)
Results of the neuropsychological tests | At inclusion (day 0)
  * Go/NoGO paradigm
  * Continuous Performance Test and virtual Continuous Performance Test
  * Stroop test and virtual stroop test
  * Wisconsin Card Sorting Test

CONTACTS AND LOCATIONS:
Overall Officials: Cyril CHAUFTON, Md, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, MD, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Bioulac S, Sagaspe P, Tron E, Benard A, Berthomier C, Brandewinder M, Philip P, Taillard J. Does Homeostatic Sleep Pressure Buildup Explain Objective Excessive Daytime Sleepiness in Adults With ADHD? An Exploratory Study. Front Psychiatry. 2021 Feb 19;12:586528. doi: 10.3389/fpsyt.2021.586528. eCollection 2021. PMID 33679469